CLINICAL TRIAL: NCT01013896
Title: Building Adherence to Live With And Navigate my CF Experience
Brief Title: Building Adherence to Live With And Navigate my Cystic Fibrosis (CF) Experience
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kristin A. Riekert, PhD, Co-Director, The Johns Hopkins Adherence Research Center, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: NA_00025417; R01HL087997-02 (NIH)
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cystic Fibrosis Education (Active Comparator): This intervention is designed to increase knowledge and enhance the skills needed to optimize CF-management. The strategies used to achieve improved adherence include providing didactic education and skills training, and proscriptively using behavioral modification strategies, such as positive reinforcement for desired behaviors, and problem-solving training to overcome barriers.
  Interventions: Other: Cystic Fibrosis Education
- Motivational Interviewing (Experimental): The Counselor's overarching goal for the intervention is to motivate and assist the participant to improve his/her adherence to the CF pulmonary medications. The intervention will begin by providing the patient personal feedback on their adherence (using pharmacy refill data) and health outcomes (e.g., trajectory of lung function values, frequency of exacerbations) as well as clinic-level figures showing the association between adherence and health outcomes.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — Among a group of older adolescents and adults with CF, we propose to evaluate the relative efficacy of a Motivational Interviewing-focused intervention (MI) in improving adherence and reducing CF-related morbidity compared to a CF education intervention (CFE; attention control group).
  Arms: Motivational Interviewing
Other: Cystic Fibrosis Education — Among a group of older adolescents and adults with CF, we propose to evaluate the relative efficacy of a Motivational Interviewing-focused intervention (MI) in improving adherence and reducing CF-related morbidity compared to a CF education intervention (CFE; attention control group).
  The Cystic Fibrosis Education serves as the attention control group.
  Arms: Cystic Fibrosis Education

SUMMARY:
The investigators research group and others have found that patient-reported adherence to all aspects of the regimen is suboptimal and objective measures suggest even poorer adherence. There is little data, however that identifies and examines the reason for nonadherence in an adult Cystic Fibrosis (CF) population or identifies effective strategies for improving adherence.

The investigators propose to evaluate the relative efficacy of a Motivational Interviewing-focused intervention (MI) in improving adherence and reducing CF-related morbidity compared to a CF education intervention (CFE; attention control group). Specifically, The investigators hypothesize that MI will result in improved regimen adherence and reduced CF morbidity compared to the CFE control group.

ELIGIBILITY:
Inclusion Criteria:

* Have a doctor confirmed diagnosis of CF
* Age 16 years old or older
* Prescribed an inhaled mucolytic, inhaled antibiotic therapy, chronic macrolide therapy and/or hypertonic saline therapy for the previous 12 months.
* Scheduled for a regular visit at either the pediatric or the adult CF clinic at Johns Hopkins Hospital.

Exclusion Criteria:

* Burkholderia cepacia complex isolated from the respiratory tract within the past 2 years.
* Had a lung transplant
* Participated in NA_00008649 A pilot study of Motivational Interviewing for adults with CF.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
A medication possession ratio (MPR) will be calculated for each prescribed drug that is being monitored for adherence. | 12 months

SECONDARY OUTCOMES:
Change in Forced Expiratory Volume in One Second (FEV1) Percent Predicted. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristin A Riekert, Ph.D., Principal Investigator — The Johns Hopkins Adherence Research Center
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States